CLINICAL TRIAL: NCT03930576
Title: Pregnancy Context and Health
Brief Title: Consequences of Unwanted Pregnancy in Nepal
Status: Active, not recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Center for Research on Environment, Health and Population Activities (Other)
Responsible Party: Sponsor
Other Study IDs: 18-25863
Record Dates: First submitted 2019-04-22; First posted 2019-04-29 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Unwanted Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Early Legal Terminations: Participants who receive a legal termination at <10 weeks gestation at a recruiting facility.
- Late Legal Terminations: Participants who receive a legal termination at 10+ weeks gestation at a recruiting facility.
- Turn-aways: Termination outside Legal Setting: Participants who receive a termination at another facility or outside the formal healthcare sector.
  Interventions: Other: Receipt of termination services outside of legal setting
- Turn-aways: Birth: Participants who ultimately carry the pregnancy to term

INTERVENTIONS:
Other: Receipt of termination services outside of legal setting — This study uses variation in gestational age to examine the impact of receipt of legal termination services compared to denial and receipt outside legal settings and birth.
  Other Names: Carrying unwanted pregnancy to term
  Groups: Turn-aways: Termination outside Legal Setting

SUMMARY:
The objective of this project is to examine the health consequences of unwanted pregnancy and denial of legal pregnancy termination services in Nepal on women and their children. The proposed study will be a large, longitudinal, prospective, quantitative study among women seeking termination services at 14 diverse facilities in 7 provinces (two facilities in each province) of Nepal. Every 6 months following baseline, surveys will cover questions about women's physical and mental health, the health and development of their children, as well as measures of family wellbeing, such as residency, relationship status and quality, and extended family relationships, and financial wellbeing, such as employment status, hours of labor, food security, income, and education.

DETAILED DESCRIPTION:
The objective of this project is to examine the health consequences of unwanted pregnancy and denial of legal pregnancy termination services in Nepal on women and their children. Births following unwanted pregnancies can be associated with negative physical, social and economic consequences for both the woman and child. Half of all unintended pregnancies are terminated before they are carried to term and, when performed in unsafe or illegal conditions, the consequences can include infection, infertility, and death. The incidence of mortality and morbidity from abortion are notoriously difficult to measure. Widespread stigma associated with unwanted pregnancy - even in settings in which termination is legally available - contribute to misreporting, concealment, and misattribution of termination-related morbidity and mortality. In addition, many women seek illegal methods-both safe and unsafe-which further confounds efforts to measure the prevalence of mortality and morbidity from terminations. The effects of unwanted pregnancy on children, including children born prior to and subsequent to the unwanted pregnancy, are also not well established. A prospective longitudinal study of women with unwanted pregnancies is required to validly investigate the health consequences for women and their families of termination outside of the legal system and delivery of an unwanted pregnancy, as compared to legal termination. Such a study is only possible in places like Nepal, where termination is legal but barriers prevent some women from receiving the service.

Aim 1: To investigate the predictors of denial of legal pregnancy termination services and identify groups of women who may be at elevated risk of adverse sequelae from unwanted pregnancy.

Aim 2: To assess the health consequences for women of childbirth and illegal termination after denial of a legal termination. By comparing the two groups of women denied termination of pregnancy to those obtaining legal procedures, the study team will assess the health effects of denial while accounting for factors associated with experience of unwanted pregnancy.

Aim 3: To measure the effects of legal and illegal termination compared to birth on the health and development of women's existing and subsequent children

Prospective longitudinal data from women in a less developed country would provide valuable evidence for the development of programs and policies globally to improve access to and utilization of safe termination services where they are legal, and harm reduction services for women who are unable to access services.

ELIGIBILITY:
Inclusion Criteria:

* women
* seeking pregnancy termination services at one of the study facilities
* self-report last menstrual period to be at least 10 weeks ago or not know her gestational age
* 15 years old or older
* live in Nepal

Exclusion Criteria:

* under 15 years old
* not pregnant
* do not live in Nepal

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: The proposed study will be a large, longitudinal, prospective, quantitative study among women seeking termination services at 14 diverse facilities in 7 provinces (two facilities in each province) of Nepal. The specific facilities were randomly selected from a list of providers who served more than 60 women in FY 2016/17. Providers who serve more than 60 women per year make up 44% of all providers but provide 92% of termination services. One non-governmental organization and one public site was randomly selected within each of 7 provinces so that their chance of selection was proportionate to the number of women served. These sites are a representative sample of women seeking care.
Sampling Method: Probability Sample
Enrollment: 1436 (Estimated)
Dates: Start 2019-04-16 (Actual); Primary Completion 2028-12-15 (Estimated); Study Completion 2028-12-15 (Estimated)

PRIMARY OUTCOMES:
Proportion experiencing denial of termination services on day of recruitment | 6 weeks
  This will be defined as the proportion of participants who did not receive termination services on the day they were recruited at the clinic site where they are recruited in to the study.
Proportion of participants who did not receive a termination from an approved facility | 6 weeks
  Proportion of participants who did not receive termination services from the recruitment clinic and did not receive a termination at any facility that they were referred to by the recruitment facility
Proportion of termination-seeking participants who received a termination | 6 months
  Participants will report their pregnancy outcome at 6 months; the proportion of participants who had an abortion by 6 months versus had a miscarriage, gave birth, or were still pregnant.
Proportion of existing children with stunting at 36 months | 36 months
  The proportion of children existing at the time of termination-seeking who having stunting, or low height-for-age, defined according to the World Health Organization as less than two standard deviations of the World Health Organization Child Growth Standards median.
Maternal deaths during the study period | 36 months
  Proportion of maternal deaths by end of study. The study team will implement a verbal autopsy protocol for any women who die during the study period, with a particular focus on identifying specific pregnancy-related causes of death.
Proportion of women reporting poor health by 36 months | 36 months
  The proportion of participants who self-report poor or very poor physical health by 36 months.
Proportion of subsequent children with stunting | 36 months
  The proportion of subsequent children born to participants after the index pregnancy who having stunting, or low height-for-age, defined according to the World Health Organization as less than two standard deviations of the World Health Organization Child Growth Standards median.

SECONDARY OUTCOMES:
Proportion experiencing violence from husband at each year of follow up | 36 months
  Proportion experiencing any physical violence from husband over time (12 months, 24 months, 36 months), defined pushed you, shake you, throw something at you (yes/no), slapped you (yes/no), twisted your arm or pulled your hair (yes/no), punched you (yes/no), kicked you (yes/no), tried to choke you (yes/no), threatened or attacked you with a weapon (yes/no).
Proportion experiencing violence from any family members or close relatives other than husband at 36 months | 36 months
  Self-reported violence from family members or close relatives other than husband or partner (yes/no) in the past 12 months.
Proportion reporting depression at 36 months | 36 months
  Proportion of participants self-reporting feeling down, depressed or hopeless nearly every day, more than half the days, or several days in the prior two weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Diana G Foster, PhD, Principal Investigator — University of California, San Francisco; Mahesh Puri, PhD, Principal Investigator — CREHPA
Locations (1):
- CREHPA, Kathmandu, Nepal

IPD SHARING:
Plan to Share IPD: No